CLINICAL TRIAL: NCT06822530
Title: PROACT: Promoting Follow-Up of Abnormal Colorectal Cancer Screening Tests Through Multilevel Interventions
Brief Title: A Multilevel Intervention to Increase Colorectal Cancer Screening Tests in Patients With Abnormal Fecal Immunochemical Test Results, PROACT Trial
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: RG1124701; NCI-2024-08639 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R37CA295618 (NIH); FHIRB0020712 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2025-01-27; First posted 2025-02-12 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Early Intervention, Educational; Educational Status; Methods; Interviews as Topic; Palliative Care

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: The program navigator will be blinded to randomization assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (usual care) (Active Comparator): Patients receive usual care from the CRC screening program navigator which includes monthly phone calls with the CRC screening program navigator, and assistance with colonoscopy scheduling.
  Interventions: Other: Best Practice; Other: Electronic Health Record Review
- Group II (usual care, video, rideshare transportation) (Experimental): Patients receive usual care as described in Group I and additionally receive a QR code with a link to a video to address patient-level fears of colonoscopy screening via text message, mailed letter, or EHR platform as well as access to transportation home after colonoscopy via a rideshare program arranged through the discharge nurse on study.
  Interventions: Other: Best Practice; Other: Educational Intervention; Other: Electronic Health Record Review; Other: Interview; Other: Supportive Care; Other: Survey Administration

INTERVENTIONS:
Other: Best Practice — Receive usual care CRC screening program navigation
  Other Names: standard of care; standard therapy
Other: Educational Intervention — Receive QR code and link to video addressing fears of colonoscopy
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Group II (usual care, video, rideshare transportation)
Other: Electronic Health Record Review — Ancillary studies
Other: Interview — Ancillary studies
  Arms: Group II (usual care, video, rideshare transportation)
Other: Supportive Care — Receive rideshare transportation home after colonoscopy
  Other Names: Supportive Therapy; Symptom Management; Therapy, Supportive
  Arms: Group II (usual care, video, rideshare transportation)
Other: Survey Administration — Ancillary studies
  Arms: Group II (usual care, video, rideshare transportation)

SUMMARY:
This clinical trial studies whether an intervention that addresses two or more levels of care (multilevel intervention) increases follow-up of abnormal, non-invasive, colorectal cancer (CRC) screening test results. The fecal immunochemical test (FIT) is a non-invasive, stool-based, CRC screening test. FITs are relatively inexpensive and can be completed at home, for these reasons, it is a preferred method of CRC screening in healthcare settings that care for under-resourced patients or have limited colonoscopy access. For FIT-based CRC screening to be effective, abnormal results must be followed by a colonoscopy, however many patients fail to complete this recommended follow-up test. The multilevel intervention addresses barriers to follow-up colonoscopy at the patient and health system levels of care through a CRC screening patient navigator, an educational video, and transportation assistance. The navigator provides patient support and assistance with colonoscopy scheduling. The educational video addresses identified patient fears around colonoscopies. Transportation assistance is offered after the colonoscopy through a rideshare program to address transportation barriers. Therefore, this multilevel intervention may increase follow-up colonoscopy completion in patients with abnormal FIT results.

DETAILED DESCRIPTION:
OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive usual care from the CRC screening program navigator which includes monthly phone calls with the CRC screening program navigator, and assistance with colonoscopy scheduling.

GROUP II: Patients receive usual care as described in Group I and additionally receive a quick response (QR) code with a link to a video to address patient-level fears of colonoscopy screening via text message, mailed letter, or EHR platform as well as access to transportation home after colonoscopy via a rideshare program arranged through the discharge nurse.

After completion of study intervention, patients are followed up for 18 months.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS: Age >= 45 years old and =< 75 years old
* PATIENTS: Receives care at an Harborview Medical Center (HMC) or University of Washington-Kent-Des Moines (UW-KDM) primary care clinic
* PATIENTS: >= 1 month from documented abnormal FIT result
* PATIENTS: Has not received a colonoscopy between the abnormal FIT and enrollment
* CLINIC STAFF: HMC or UW-KDM physician or staff member who provides primary care or gastroenterology care
* CLINIC STAFF: Staff in the Fred Hutchinson (Fred Hutch)/UW Medicine Population Health Program that provide colorectal cancer screening and navigation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 682 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Rate of colonoscopy completion within 6 months | At 6 months after randomization
  Will descriptively compare the rates of colonoscopy completion at 6 months. Will fit a generalized mixed effects model with a logit link and a random effect for clinic. Will include an indicator variable for the randomized group (usual care versus (vs.) multilevel intervention) and adjust for patient-level clinical and demographic factors (e.g., age, sex, race, ethnicity, primary language, marital status, last primary care visit, insurance) and clinic-level factors (e.g., clinic size, average full-time equivalent providers per clinic, average provider panel size, primary care provider mix (Doctor of Medicine/Doctor of Osteopathic Medicine vs. other advanced degree).
Time to colonoscopy completion | Beginning 6 months after randomization until study completion
  Will assess the time to colonoscopy completion in days and compare these times across individual clinics.

SECONDARY OUTCOMES:
Rate of colonoscopy completion > 6 months | At 9 and 12 months after randomization
  Will fit separate generalized mixed effects model for each binary outcome, with a logit link and a random effect for clinic. In all models, will include an indicator variable for the randomized group and adjust for patient-level clinical and demographic factors and clinic-level factors.
Colonoscopy referral: Number of participants referred for a colonoscopy | Up to 18 months after randomization
  Will assess colonoscopy referral (yes/no) as the number of participants who have a colonoscopy referral placed after randomization.
Time to colonoscopy referral (days) | Up to 18 months after randomization
  Will assess the number of days from randomization to colonoscopy referral.
Number of participants who schedule a colonoscopy | Up to 18 months after randomization
  Will assess the number of referred participants who schedule a colonoscopy.
Time to scheduling a colonoscopy (days) | Up to 18 months after randomization
  Will assess the number of days from randomization to a colonoscopy being scheduled.
Time from abnormal fecal immunochemical test (FIT) result to colonoscopy completion | Up to 18 months after randomization
  Will assess the time from abnormal FIT results to colonoscopy completion (days). Will fit separate generalized mixed effects model for each binary outcome, with a logit link and a random effect for clinic. For time-to-event secondary outcomes, will fit separate Cox proportional hazards regression models where the outcomes will be measured in days. In all models, will include an indicator variable for the randomized group and adjust for patient-level clinical and demographic factors and clinic-level factors.
Rates of colorectal cancer or advanced adenoma | Up to 18 months after randomization
  Will assess the number of colorectal cancers or advanced adenomas detected as reported in pathology reports. Colorectal cancer will be defined as a histologically confirmed invasive carcinoma or minimally invasive carcinoma. Advanced adenoma will be defined as a tubular adenoma > or = 10mm, villous, or high-grade dysplasia.
Proportion and demographic characteristics of individuals who are eligible and receive the multilevel intervention after randomization (Reach) | 6-24 months post randomization
  Participant demographics and quantitative measures of implementation outcomes (reach) will be reported as proportions or medians and interquartile ranges (IQRs). Average scores of the implementation outcomes will be reported per participant and clinic. Will assess differences between groups using chi-square, Student's t-test or Wilcoxon tests, as appropriate.
Perception that the intervention components are suitable to address identified barriers (Acceptability) | 6-24 months post randomization
  Participant demographics and quantitative measures of implementation outcomes (acceptability) will be reported as proportions or medians and IQRs. Average scores of the implementation outcomes will be reported per participant and clinic. Will assess differences between groups using chi-square, Student's t-test or Wilcoxon tests, as appropriate. Semi-structured interviews will be transcribed verbatim, verified against recordings, and uploaded to the data management software by participant number. Will apply a hybrid approach to the data analysis by combining inductive and deductive methods. Using a convergent parallel mixed-methods approach, will integrate and analyze quantitative and qualitative data, according to the Predisposing, Reinforcing, and Enabling Constructs in Educational Diagnosis and Evaluation model that analyzes data at multiple ecological levels and is particularly relevant for the study.
Degree to which the intervention is used as intended (Fidelity) | 6-24 months post randomization
  Will be assessed by the proportion and demographic characteristics of individuals who use all components of the intervention after randomization, complete adherence to the program protocol, and quality of the program delivery. Participant demographics and quantitative measures of implementation outcomes (fidelity) will be reported as proportions or medians and IQRs. Average scores of the implementation outcomes will be reported per participant and clinic. Will assess differences between groups using chi-square, Student's t-test or Wilcoxon tests, as appropriate.
Average cost per patient to deliver the intervention | Weekly, for up to 8 months
  Will calculate personnel and operational costs for the multilevel intervention for each patient. Total costs for each component per patient (personnel, materials/supplies, facility fees, training, and professional development) will also be calculated.
Average cost per clinic to deliver the intervention | Weekly, for up to 8 months
  Will calculate personnel and operational costs for the multilevel intervention for each clinic. Total costs for each component per clinic (personnel, materials/supplies, facility fees, training, and professional development) will also be calculated.
Proportion of costs per intervention activity | Weekly, for up to 8 months
  Will calculate the proportion of costs that can be attributed to each intervention activity.
Number of participants served per intervention component | Weekly, for up to 8 months
  The number of participants served per intervention component.
Average cost per participant by intervention component | Weekly, for up to 8 months
  Will calculate an average per-participant activity cost for each intervention component.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel B. Issaka, MD, MAS, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD to be shared with other researchers: All of the IPD collected during the trial, after deidentification. Supporting information that will be shared will include: Study protocol, analyzable data set, data dictionary/codebook, statistical analysis plan, analytic code, data collection instruments.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Complete trial data will be made available no later than 12 months via clinicaltrials.gov after the trial's primary completion date regardless of whether the clinical trial was completed as planned or terminated earlier in compliance with the NCI Clinical Trial Access Policy. Participant data, interview transcripts and underlying primary data for the publications will be made available through Mendeley data repository no later than the time of an associated publication or the end of the performance period, whichever comes first. Data will remain available via Mendeley indefinitely.
Access Criteria: Public-access data will be available to researchers through the Mendeley website. IPD will be made available to researchers who provide a methodologically sound proposal to achieve the aims in their proposal and obtain approval from an independent review committee. Researchers who wish to use the most sensitive data and/or link project data to other datasets must apply for access through a contract request to use the Mendeley virtual data enclave.
URL: https://data.mendeley.com/